CLINICAL TRIAL: NCT03422926
Title: ChildObesity180 - Social Marketing Campaign to Encourage Healthful Eating in Restaurants for Children
Acronym: CO180
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PV1529
Record Dates: First submitted 2017-04-24; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Child Overnutrition
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Social marketing messaging campaign
  Interventions: Behavioral: Social marketing campaign
- Control (No Intervention): No messaging campaign

INTERVENTIONS:
Behavioral: Social marketing campaign — Messaging campaign designed to help mothers in choosing healthful options when dining out.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether a messaging campaign affects the calories ordered for and consumed by children in a quick serve restaurant setting.

DETAILED DESCRIPTION:
ChildObesity180 seeks to develop and implement a messaging campaign informed by evidence-based behavioral theory as well as perspectives from parents, children, and the restaurant industry. The campaign aims to help parents choose healthful options for their children when dining in the quick-serve restaurant setting. Aim 1 is campaign development. Aims 2 and 3 are assessment (i.e., Randomized controlled trial and revenue analysis). Hypotheses are that the messaging campaign will be associated with fewer calories ordered/consumed by children in the quick serve setting; and the campaign will not negatively impact quick serve restaurant revenue.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of a 4 - 12 year old child (who is present)
* Have not participated in the study before
* <<Intervention community only>> live, work, or frequently travel to community

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2646 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
kilocalories ordered | change from baseline to follow-up 3-5 months later
  Receipt data will be used to determine what items were ordered for the parent and child, and kcals will be calculated using nutrition information from the restaurant and bomb calorimetry.
kilocalories consumed | change from baseline to follow-up 3-5 months later
  Child plate waste will be collected, weighed and digitally imaged; a subset will be analyzed using bomb calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Christina D Economos, PhD, Principal Investigator — Tufts University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hennessy E, Shonkoff E, Harelick L, Bakun P, Chui K, Roberts S, Folta S, Goldberg J, Economos CD. The impact of a community social marketing campaign on children's meal orders and consumption: main outcomes from a group randomised controlled trial. Public Health Nutr. 2023 Jan;26(1):256-261. doi: 10.1017/S136898002200163X. Epub 2022 Aug 8. PMID 35938500